CLINICAL TRIAL: NCT04323371
Title: Cardiogenic Shock Integrated PHenotyping for Event Reduction
Acronym: CIPHER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 43-12022020
Record Dates: First submitted 2020-03-11; First posted 2020-03-26 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure
Keywords: heart failure; cardiogenic shock; endothelial glycocalyx; Angiopoietin (Ang)-2; Metabolomics
MeSH Terms: conditions — Heart Failure; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples (blood and derived fluids)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute decompensated heart failure: patients admitted with Acute decompensated heart failure Complicated by cardiogenic shock
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Diagnostic Test: ELISA — Blood and derived fluids will be collected from 26 ADHF CS patients admitted to intensive care at Niguarda Hospital and locally stored.Stocked samples will be shipped to the Central Laboratories at Milano Uni and MilaIFC-CNR for the metabolomic and biomarkers analysis,respectively.To evaluate interleukin-6 (marker of systemic inflammation),angiopoietin-2 (marker of endothelial permeability), syndecan-1 and heparan sulfate (markers of endothelial glycocalyx),2 aliquotes of serum samples will be used by IFC CNR.The biomarkers will be assessed through ELISA analytical techniques, based on the interactions inside a microplate between a primary pre-coated antibody and the specific protein contained in serum samples.A secondary antibody, link to a horseradish peroxidase (HRP) detection system, is able to recognize and bind the antigen, and to produce a colorimetric reaction after the addition of enzyme substrate which is proportional to the amount of the target protein bound

SUMMARY:
The purpose of this study is to better understand the time course of different biological mechanisms involved in acute decompensated heart failure complicated by cardiogenic shock throughout the evaluation of changes and the relationship among markers of inflammation (IL-6) and markers of increased endothelial permeability (Ang-2) or endothelial glycocalyx perturbation (Syndecan-1 and HS) and throughout a targeted metabolomic approach.

DETAILED DESCRIPTION:
Cardiogenic shock (CS) is a heterogenous syndrome with in-hospital mortality up to 60%, that, unfortunately, has remained stagnant over the time, despite observed improvements with pharmacological and non-pharmacological approach, even though only in terms of haemodynamic stabilization.

While very early mortality in CS is largely related to sudden and severe circulation failure, subsequent death is strongly influenced by activation of neurohumoral and inflammatory response leading to multiorgan failure. Previous studies on CS have almost exclusively been focused on CS following an acute coronary syndrome (ACS). Patients with acutely decompensated heart failure (ADHF) represent a different pathophysiologic phenotype compared with acute coronary syndrome (ACS) patients, which may lead to a differential response to device therapy.

In the face of complex biological phenomena guidelines are incapable of distinguishing the underlying pathophysiological mechanisms and give us input to standardize, whereas there is an unmet need for a personalized medicine.

The evaluation of changes and the relationship among markers of inflammation (IL-6) and markers of increased endothelial permeability (Ang-2) or endothelial glycocalyx perturbation (Syndecan-1 and HS) and an exploratory analysis throughout targeted metabolomics may help us to better understand the time course of different biological mechanisms involved in CS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and < 75, men and women;
* 1) Systolic blood pressure (SBP) < 90mmHg or mean arterial pressure (MAP) < 60 mmHg, after an appropriate fluid challenge if there is no sign of overt fluid overload; OR 2) need of vasoactive agents to maintain SBP > 90 mmHg or MAP > 60 mmHg.
* Reduced ejection fraction (left ventricle systolic function ≤35%).
* Moreover, eligible patients have to fit at least ONE of the following criteria/items of overt hypoperfusion: altered state of consciousness; sweaty and cold skin; mixed venous oxygen saturation < 60%; arterial lactates > 2 mmol/L; oliguria < 0.5 ml/Kg/h for at least 6 hours.
* Eligible patients shouldn't have contraindications to heart replacement therapy (HRT).

Exclusion Criteria:

The participant will not be enrolled if ANY of the following criteria will be detected:

* Cardiogenic shock symptoms beyond 6 hours.
* Septic shock with evident septic focus.
* Cardiogenic shock due to acute myocardial infarction.
* Cardiogenic shock due to acute myocarditis.
* Cardiogenic shock due to pulmonary thromboembolism.
* Reiterating major arrhythmias: VT or VF or AF, with ventricular rate > 160 bpm.
* Severe aortic valve disease.
* Obstructive hypertrophic cardiomyopathy or constrictive pericarditis or severe heart failure due to congenital heart disease
* Severe peripheral vascular disease that contraindicates mechanical support insertion.
* Cardiogenic shock secondary to either cardiac or non-cardiac surgery.
* Comorbidities with ominous prognosis (life expectancy < 1 year).
* Estimated glomerular filtration rate severely impaired before enrolment (eGFR<30 ml/min/1.73 m2) or severe chronic obstructive pulmonary disease (COPD) or liver cirrhosis.
* Pregnant, lactating or subjects planning pregnancy during the course of the trial.

Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 18 Years to 74 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with acute decompensated heart failure, complicated by cardiogenic shock
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Value of Interleukin 6 (IL-6) | 3 years
  Markers of inflammation. Unit of measure: pg/mL.
Value of Angiopoietin 2 (Ang-2) | 3 years
  Markers of endothelial permeability. Unit of measure: ng/mL.
Value of Syndecan-1 | 3 years
  Endothelial glycocalyx perturbation. Unit of measure: ng/mL.
Value of Heparan sulfate (HS) | 3 years
  Endothelial glycocalyx perturbation: Unit of measure: ug/mL.
Metabolomics profiling | 3 years
  Exporatory assessment of targeted metabolomics through the quantification of almost 180 molecules, including acylcarnitines, amino acids and biogenic amines, hexoside, sphingolipids and glycerophospholipids.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided